CLINICAL TRIAL: NCT07296224
Title: Scannographic Predictive Factors of Changes in the Intraoperative Therapeutic Strategies During Metabolic Bariatric Surgery (MBS)
Brief Title: Scannographic Predictive Factors of Change of Strategy During Metabolic Bariatric Surgery
Acronym: SCANOBE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, NOMINE-CRIQUI Claire, MD Head of endocrine surgery Unit, Central Hospital, Nancy, France
Other Study IDs: FORM-03935
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
Keywords: metabolic bariatric surgery; obesity; gastric bypass; sleeve
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent a change of surgical strategy: patients who underwent an other surgical strategy than gastric by pass : laparoscopic sleeve gastrectomy, sleeve gastrectomy or gastric bypass by laparotomy, no metabolic bariatric surgery (procedure impossible to achieve)
- control group: patients who underwent laparoscopic gastric bypass. Each patient who had undergone a change in strategy was subsequently randomly matched with three 'controls' who were comparable in terms of age (within 5 years of each other), sex and body mass index (BMI). The controls were defined as patients with the same inclusion criteria as those patients in the 'change of strategy' group

SUMMARY:
Background: Laparoscopic Roux-en-Y Gastric By-pass (LRYGB) is not always feasible due to intraoperative difficulties, necessitating a change during surgical procedure. Non-contrast abdominal CT scans is not recommended before bariatric surgery but could be informative and very few studies have evaluated the relevance of these scans. The primary objective was to identify CT scan criteria that could predict a change in the intraoperative therapeutic strategy during LRYGB. Secondary objectives included identifying clinical data associated with change of intraoperative strategy, the impact of surgeon's experience and evaluate postoperative complications.

Methods: The study was conducted in University Hospital of Nancy, France between October 2012 and December 2022. This retrospective matched-case-control study (1:3) compared patients with intraoperative change of strategy when LRYGB was initially planned (study group) versus matched patients who undergone LRYGB. Clinical, scannographic, surgical experience and postoperative complications data were collected in the two groups.

DETAILED DESCRIPTION:
Obesity is a multifactorial condition involving behavioral, environmental and genetic factors . Possible treatments for obesity include nutritional, dietary and cognitive-behavioral management, as well as pharmacological therapies and metabolic bariatric surgery (MBS) . These treatments must be combined and tailored to each patient.

Before the performance of MBS only an esogastroduodenal endoscopy with systematic biopsies for Helicobacter pylori is currently recommended . In France, abdominal ultrasound is added for detecting vesicular lithiasis . According to the American Society for Metabolic and Bariatric Surgery abdominal ultrasound is indicated in patients presenting biliary tract symptoms or liver disease . Non-contrast abdominal CT scan is not an aspect of the initial assessment in Europe or in the United States . To our knowledge, only one MBS team evaluated the value of preoperative CT scans for identifying silent pathologies and concluded that the value of CT scans were minimal . In Nancy University Hospital, a preoperative non-contrast abdominal CT scan is proposed to all patients scheduled for MBS to screen for incidental lesions, hiatal hernia not visible in endoscopy and left liver hypertrophy.

In Nancy University Hospital, a Laparoscopic Roux-en-Y gastric bypass (LRYGB) is preferentially performed. Due to surgical difficulties, LRYGB is not always an option for treatment. In these cases, a change in the surgical procedure may be needed. In very difficult cases, the performance of any MBS may be impossible.

The investigator hypothesizes that preoperative scannographic features-especially increased left liver volume (LLV) -are predictive of intraoperative strategy change during LRYGB, and that this risk is further influenced by patient history and surgeon experience.

Design This was a retrospective, single-center, observational case-control study conducted between 1st October 2012 and 31st December 2022 at the University Hospital of Nancy.

Population All adult patients scheduled for LRYGB surgery at the Nancy University Hospital between 1st October 2012 and 31st December 2022 who underwent a change in intraoperative surgical strategy and who did not object to the collection of their data were identified. Patients who did not have a preoperative scan and those who were lost to follow-up within 6 months of surgery were excluded.

Based on surgical reports, a change in surgical strategy was defined as follows: patients who underwent laparoscopic sleeve gastrectomy, laparotomy Roux-en-Y gastric bypass or laparotomy sleeve gastrectomy instead of a LRYGB and patients who experienced an interruption of the procedure during LRYGB.

Each patient who had undergone a change in strategy was subsequently randomly matched with three 'controls' who were comparable in terms of age (within 5 years of each other), sex and body mass index (BMI). The controls were defined as patients with the same inclusion criteria as those patients in the 'change of strategy' group but who had undergone a LRYGB.

Collected data The clinical data that were collected included age, sex, weight, height, BMI, history of abdominal surgery, hypertension, diabetes, obstructive sleep apnoea syndrome, non-alcoholic fatty liver disease and dyslipidemia. Surgeon's experience reported as junior (≤100 cases of MBS) or senior (>100 cases of MBS), A unique radiologist who was unaware of the patient's details and surgical history analysed preoperative non-contrast abdominal CT scans and used Aw Server version 3.2. The preoperative scan criteria included parietal thickness, the peritoneal height/width ratio in axial section and the visceral perimeter at L1, the umbilical perimeter, the total psoas area (TPA) (mm2) at L3 and the LLV . The measurement of visceral perimeter, umbilical perimeter and total psoas area was performed using manual measurement. The measurement of the LLV was performed using semi-automatic measurement adjusted by the radiologist as necessary.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for LRYGB surgery at the Nancy University Hospital between 1st October 2012 and 31st December 2022 who underwent a change in intraoperative surgical strategy
* patient who did not object to the collection of their data.
* patients over the age of 18

Exclusion Criteria:

* Patients who did not have a preoperative scan
* patients who were lost to follow-up within 6 months of surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients scheduled for LRYGB surgery at the Nancy University Hospital between 1st October 2012 and 31st December 2022.
  Patients with body mass index > 35 kg/m2 selected to underwent bariatric surgery by the medical and surgical team Patients with preoperative CT scan
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
left liver volume scannographic measure | between 1st October 2012 and 31st December 2022
  the Left Liver Volume (LLV) was measured on an abdominal CT scan by a raidologist

SECONDARY OUTCOMES:
parietal thickness | between 1st October 2012 and 31st December 2022
  parietal thickness was measured on abdominal CT scan
surgical experience, number of bariatric procedure done before the surgery studied (less than 100 procedures or more) | between 1st October 2012 and 31st December 2022
  Surgeon's experience reported as junior (≤100 cases of MBS) or senior (>100 cases of MBS)
Post operative morbidity | between 1st October 2012 and 30st June 2023
  Post-operative morbidity was evaluated using Clavien-Dindo classification ,180 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nancy, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: Undecided